CLINICAL TRIAL: NCT02852343
Title: Etude de Concordance Entre la Technique OSNA et Les Techniques Classiques Pour la Recherche de métastases Ganglionnaires Des Cancers Des VADS
Brief Title: One-step Nucleic Acid Amplification for Detecting Lymph Node Metastasis of Head and Neck Squamous Cell Carcinoma
Acronym: OSNA-ORL
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC14_9878
Record Dates: First submitted 2016-07-19; First posted 2016-08-02 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: cN0 Oral Squamous Cell Carcinomas

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The investigators main objective is to show that OSNA technique is as accurate as pathological analysis (frozen section / HE staining and immunochemistry) to detect occult lymph node metastasis (micro and macrometastasis).

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years old
* Head and neck squamous cell carcinoma diagnosed by biopsy
* N0 classification (N0: no lymph node invasion on clinical and radiological examination).
* Neck dissection or sentinel lymph node biopsy required to treat the patient
* ECOG 1,2 or 3
* Patient's consent

Exclusion Criteria:

* Patient previously treated by radiotherapy or surgery for head and neck neoplasm.
* Contraindication or patient unwillingness to undergo surgical treatment
* Incapacitated adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with sceduled procedure to cN0 oral squamous cell carcinomas
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2015-01-05 (Actual); Primary Completion 2016-12-21 (Actual); Study Completion 2016-12-21 (Actual)

PRIMARY OUTCOMES:
number of CK19 mRNA copies/µL of diluted lymph node lysate | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier universitaire de Rennes, Rennes, France

REFERENCES:
- [Derived] Peigne L, Godey F, Le Gallo M, Le Gall F, Fautrel A, Morcet J, Jegoux F. One-step nucleic acid amplification for detecting lymph node metastasis of head and neck squamous cell carcinoma. Oral Oncol. 2020 Mar;102:104553. doi: 10.1016/j.oraloncology.2019.104553. Epub 2020 Jan 28. PMID 32004908